CLINICAL TRIAL: NCT05243160
Title: Implementing Medication Reviews Through Interdisciplinary Dialogue in Patients With Coexisting Diabetes and Mental Illness
Brief Title: Medication Reviews in Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Collaborators: Steno Diabetes Center Sjaelland (Other Government); Region Zealand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PRURegionZealand18
Record Dates: First submitted 2022-01-17; First posted 2022-02-16 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia; Diabetes; Metabolic Syndrome; Severe Mental Disorder; Major Depressive Disorder; Bipolar Disorder; Psychosis; Psychotic Disorders
Keywords: polypharmacy; medication review; metabolic disorder; drug interaction; pharmacologist/ or clinical pharmacology/ or pharmacology/; drug interaction/; adverse drug reaction/; side effect; medication therapy management/; pharmacovigilance/; severe mental illness
MeSH Terms: conditions — Schizophrenia; Diabetes Mellitus; Metabolic Syndrome; Mental Disorders; Depressive Disorder, Major; Bipolar Disorder; Psychotic Disorders; Metabolic Diseases; Drug-Related Side Effects and Adverse Reactions | interventions — Medication Review

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Treatment as usual
- Intervention (Experimental): Intervention group will be exposed to a medication review by a clinical pharmacologist
  Interventions: Other: medication review

INTERVENTIONS:
Other: medication review — The intervention consist of a medication review by a clinical pharmacologist.
  Arms: Intervention

SUMMARY:
This study aims to investigate the potential beneficial effects of a medication review by a clinical pharmacologist on patients with coexisting severe mental illness and diabetes. The study is an intervention study in which an intervention group is assigned to the medication review whereas a control group is not. Both groups are tested using an extensive test battery at baseline and 6 months after inclusion.

Furthermore a qualitative data assessment will be undertaken using interviews and/or surveys in order to show any obstacles in implementing the intervention. This is relevant as medication reviews, performed by clinical pharmacologists as well as pharmacists, are not always implemented by the primary physician.

The economic impact of the medication review will furthermore be assessed.

DETAILED DESCRIPTION:
The effects of a medication review on patients with coexisting severe mental illness and diabetes:

Introduction:

Severe mental illness (SMI) is associated with an increased risk of diabetes (DM) and metabolic complications. The risk of type-2 diabetes is increased 2-3 fold in patients with SMI compared to the average population. This may lead to polypharmacy hence adverse drug interactions as well as adverse side effects emphasizing the need for a thorough medication review. Medication reviews by pharmacists is widely used and implemented in clinical practice. However, to the investigators knowledge studies on medication reviews by medical doctors specialized in the field of clinical pharmacology let alone on this patient cohort is scarce. Hence, this study seeks to investigate the effects of a medication review by a clinical pharmacologist on patients with coexisting severe mentall illness and diabetes.

Quality control:

The study protocol will be send for approval by the Danish National Committee on Health Research Ethics. Regarding data managing the study is send to Region Zealand's list of ongoing projects thereby ensuring responsible data managing in accordance with the current legislation.

Randomization:

The investigators aim to enroll approximatively 50 patients suffering from both severe mentall illness and diabetes (all types) in this study. Patients are drafted from the fusion clinic in Slagelse Denmark. The fusion clinic is a novel collaboration between endocrinologists and psychiatrists based in Slagelse Hospital department of psychiatry caring for patients with mental illness and diabetes. The clinic seeks to unite endocrinologists and psychiatrists in order to provide the best possible care for patients with coexisting severe mental illness and diabetes. Patients enrolled at the fusion clinic is invited to participate in this study and after having read and accepted the terms as well as the conditions of the study patients will be randomized to an intervention group as well as a control group. Using block-randomization patients will be distributed in blocks (3:3) thereby preventing any carry-over effect. Treatment arm allocation is hidden from the investigator thereby improving the quality of the data.

Data management:

Data will be accessible for co-authors as well as co-investigators participating in this study. Data will be entered into the RedCap module and written consent forms will be uploaded to this platform. Written files will be stored for 5 years at a safe location according to current legislation.

Intervention:

At baseline all participants recruited will undergo the following ratings: PANSS-6 (positive and negative syndrome scale), "UKU side effects rating scale" a danish acronym for the "Task force for clinical investigations- rating scale" a rating scale for measuring side effects associated with psychopharmacological treatment, MARS (medication adherence rating scale), CGI (clinical global impression scale), Hamilton-rating scale, Young manic rating scale and SF-12 (short form survey). Furthermore, data on medicinal load, potential drug-interactions, as well as potential side effects will be obtained at baseline. The intervention group will then be subject to a medication review by a clinical pharmacologist at the beginning of the trial whereas the control group will not. 6 months after the inclusion date both groups will be subject to the same test battery thereby showing any potential differences between the two groups.

Furthermore a qualitative data assessment of the intervention will be included in this study by interviewing clinicians and their percieved experience in using the medication review. The qualitative assessment will help to illuminate potential obstacles or barriers in implementing the medication review in real clinical practice.

Recruitment:

All patients will have to accept a written consent form thereby agreeing to participate in this study. By giving consent, the participant gives the examiner access to the patient record hence health data regarding the participant. Patients are at any time able to withdraw their consent throughout the study without effecting their ongoing treatment.

Ethics:

At the end of the study trial all patients will be offered the medication review thereby ensuring that all patients benefit from this additional expert assessment. The trial does not interfere with the usual treatment and there seems to be no additional risks for the patients participating in this study.

Funding:

The study is funded by the Steno diabetes center region Zealand Denmark and contains enough funding for 1 year of research. The research group is in the process of applying for funding for a 3- year research employment (ph.d.).

Perspective:

The investigators speculate as to whether a medication review by a clinical pharmacologist can improve not only the medicinal load but also reduce side effects, minimize adverse drug interactions, reduce financial burden asscoiated with the pharmacological treatment as well as manifest in a clinical difference for the patients. If the intervention proves useful the medication review is easily implemented in the Danish clinical practice and is therefore of relevance for the clinicians.

ELIGIBILITY:
Inclusion Criteria:

* The patients drafted must have diabetes (unspecified) and severe mental illness in this case schizophrenia, severe ADHD, anxiety, any other psychotic disorders or an affective disorder (e.g. bipolar disease and major depression). Patients are drafted from the "fusion clinic" in Slagelse Denmark which is a collaboration between endocrinologists and psychiatrists in the joint treatment of patients with diabetes and mental illness.
* Only adult patients

Exclusion Criteria:

* none of the above
* Pediatric patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Medicinal load | 6 months
  Total amount of drugs prescribed
Adverse drug interactions | 6 months
  Amount of potential drug interactions
Adverse side effects | 6 months
  The number of potentiel drug related side effects

SECONDARY OUTCOMES:
UKU side effect rating scale ("UKU" is a danish acronym for the "Task force for clinical investigations") | 6 months
  Measuring side effects related to psychopharmacological treatment. Score ranges from 0 to 54 as the maximum score. High scores corresponding to an increased burden of side effects
SF-12 (short form survey) | 6 months
  Changes in the SF-12 scale during study period. Score ranges from 0 to 100 with 100 as maximum. High scores illustrating a percieved sense of good health.
MARS (medication adherence rating scale). | 6 months
  Measuring adherence to pharmacological treatment. Score ranges from 0 to 10 with 10 as maximum value. Increased score illustrating poor adherence to the pharmacological treatment.
CGI (Clinical Global impression scale) | 6 months
  Clinical Global impression scale: Score ranges from 1-7 with increasing score illustrating poor clinical status: Higher scores corresponding to the severity of the illness.
PANSS-6 (positive and negative syndrome scale) | 6 months
  Changes in the PANSS-6 scale during study period. Scores ranges from 7-42 with increasing score as illustrating the severity of symptoms
Hamilton-17 | 6 months
  Rating scale used in rating depressive disorders. Scores rating from 0-52 with increasing score as indication of disease severity
Young manic rating scale (YMRS) | 6 months
  Rating scale used for rating bipolar episodes. Scores rating from 0-56 with increasing score as indication of disease severity
Biomarkers | 6 months
  Relevant biochemical tests related to psychotropic treatment (e.g. low density lipoprotein, high density lipoprotein, hemoglobin 1 Ac (Hb1Ac) and triglycerides).

CONTACTS AND LOCATIONS:
Overall Officials: Gesche Jürgens, MD, Study Director — Consultant physician
Locations (1):
- Research Unit for Psychotherapy and Psychopathology, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: No